CLINICAL TRIAL: NCT00207727
Title: A Phase II, Double-blind, Placebo-Controlled, Randomized, Dose-ranging Study of Multiple Subcutaneous Injections of Human Monoclonal Antibody to IL-12p40(CNTO1275) in Subjects With Relapsing-remitting Multiple Sclerosis
Brief Title: A Safety and Efficacy Study of CNTO1275 in Patients With Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Collaborators: Centocor BV (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR005284
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2009-12-02 (Estimated); Last update posted 2012-04-23 (Estimated); Status verified 2012-04

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Ustekinumab

INTERVENTIONS:
Drug: CNTO 1275

SUMMARY:
The purpose of the study is to evaluate the effectiveness and safety of CNTO 1275 in patients with Multiple Sclerosis

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a life-long disease that usually starts in young adults. In MS, inflammation and damage to nerve cells occur in the brain and spinal cord. Symptoms of MS are quite variable and may range from being mild to severe and from short to long lasting. People with MS may have a wide variety of symptoms ranging from mild to disabling. Some of thesymptoms of MS include visual disturbances such as double vision, weakness in arms or legs,difficulty with coordination, fatigue, changes in sensations such as numbness and tingling, or difficulties with concentration or memory.The drug being tested in this research study is an antibody called CNTO 1275. Antibodies are natural substances made by the body that stick to and react with other substances in the body that may cause diseases. The body makes antibodies mainly to fight infections. CNTO 1275 is an antibody that has been manufactured in the laboratory. In the test tube, CNTO 1275 sticks to and blocks the activity of a naturally occurring substance in the body called interleukin 12 (IL-12).Higher than normal levels of IL-12 have been found in people who have MS. CNTO 1275 has been tested in animals with a condition similar to MS. In those animals, IL-12 was over-produced.Animals treated with CNTO 1275 showed decreased symptoms of the condition.The purpose of this study is to better understand the safety and effectiveness of CNTO 1275 in people who have relapsing-remitting MS

Patients will receive subcutaneous injections of 30, 100, 200 mg of CNTO 1275 or placebo at Weeks 0, 1, 2, 3, 7, 11, 15, and 19 or 100 mgs at weeks 0,1,2,3,11 and 19 and placebo at wks 7 and 15.

ELIGIBILITY:
Inclusion Criteria:

* Have a definite diagnosis of Relapsing remitting Multiple Sclerosis
* Have a history of at least 1 of the following:a. A minimum of 2 relapses of MS within the previous 2 years but not within the 1-month period prior to screening. b. A relapse of MS within the previous 6 months but not within the 1-monthperiod prior to screening

Exclusion Criteria:

* Have a CNS disease (eg, CNS lymphoma, systemic lupus erythematous)
* Have significant bulbar involvement of MS or other neurologic deficits
* Have a decubitus ulcer
* Have received immunomodulatory therapies within 3 months of screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2004-07; Primary Completion 2006-03 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.

REFERENCES:
- [Derived] Robinson D Jr, Zhao N, Gathany T, Kim LL, Cella D, Revicki D. Health perceptions and clinical characteristics of relapsing-remitting multiple sclerosis patients: baseline data from an international clinical trial. Curr Med Res Opin. 2009 May;25(5):1121-30. doi: 10.1185/03007990902797675. PMID 19317608
- [Derived] Segal BM, Constantinescu CS, Raychaudhuri A, Kim L, Fidelus-Gort R, Kasper LH; Ustekinumab MS Investigators. Repeated subcutaneous injections of IL12/23 p40 neutralising antibody, ustekinumab, in patients with relapsing-remitting multiple sclerosis: a phase II, double-blind, placebo-controlled, randomised, dose-ranging study. Lancet Neurol. 2008 Sep;7(9):796-804. doi: 10.1016/S1474-4422(08)70173-X. PMID 18703004

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 249 patients were enrolled in the trial to receive either placebo or ustekinumab (CNTO 1275). There were 38 investigative sites in North America, Europe and Australia.
Groups:
- Group I: Placebo: Patients received Placebo subcutaneous (SC) injection(s) at Weeks 0, 1, 2, 3, 7, 11, 15, and 19
- Group II: Ustekinumab 27 mg Every 4 Weeks: Patients received 27 mg ustekinumab SC injection at Weeks 0, 1, 2, 3, 7, 11, 15, and 19.
- Group III: Ustekinumab 90 mg Every 8 Weeks: Patients received 90 mg ustekinumab SC injection at Weeks 0, 1, 2, 3, 11, and 19. Placebo SC injection at Weeks 7 and 15.
- Group IV: Ustekinumab 90 mg Every 4 Weeks: Patients received 90 mg ustekinumab SC injection at Weeks 0, 1, 2, 3, 7, 11, 15, and 19.
- Group V: Ustekinumab 180 mg Every 4 Weeks: Patients received 180 mg ustekinumab SC injections at Weeks 0, 1, 2, 3, 7, 11, 15, and 19.
Period: Overall Study
Arm/Group | Group I: Placebo | Group II: Ustekinumab 27 mg Every 4 Weeks | Group III: Ustekinumab 90 mg Every 8 Weeks | Group IV: Ustekinumab 90 mg Every 4 Weeks | Group V: Ustekinumab 180 mg Every 4 Weeks
Started | 49 | 50 | 50 | 50 | 50
Completed | 11 | 8 | 9 | 13 | 16
Not Completed | 38 | 42 | 41 | 37 | 34
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0
Not completed — Other | 38 | 41 | 41 | 37 | 33

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I: Placebo | Group II: Ustekinumab 27 mg Every 4 Weeks | Group III: Ustekinumab 90 mg Every 8 Weeks | Group IV: Ustekinumab 90 mg Every 4 Weeks | Group V: Ustekinumab 180 mg Every 4 Weeks | Total
Number analyzed (Participants) | 49 | 50 | 50 | 50 | 50 | 249
Age Continuous [Mean (Standard Deviation); unit: Years] | 36.3 (10.65) | 39.0 (10.34) | 38.6 (11.53) | 39.8 (11.01) | 41.1 (8.34) | 39.0 (10.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 32 | 37 | 33 | 36 | 175
  Male | 12 | 18 | 13 | 17 | 14 | 74

OUTCOME MEASURES:

1. Primary Outcome: The Cumulative Number of Newly Gadolinium-enhancing T1-weighted Lesions on Cranial Magnetic Resonance Imaging (MRI)s Through Week 23.
Description: A newly Gadolinium (Gd) enhancing T1-weighted lesion is defined as a lesion that is enhanced on a current cranial MRI scan but was not classified as a newly Gd enhancing T1-weighted lesion on the previous MRI scan.
Time Frame: Week 23
Population: Intent to treat. Missing data was imputed. The average number of newly Gd enhancing T1-weighted lesions from all valid visits for the patient will be used when prohibited medications are initiated.
Measure: Median (Inter-Quartile Range); unit: Lesions
Arm/Group | Group I: Placebo | Group II: Ustekinumab 27 mg Every 4 Weeks | Group III: Ustekinumab 90 mg Every 8 Weeks | Group IV: Ustekinumab 90 mg Every 4 Weeks | Group V: Ustekinumab 180 mg Every 4 Weeks
Number analyzed (Participants) | 49 | 50 | 50 | 50 | 50
Lesions | 1.20 [0.00 to 9.60] | 1.00 [0.00 to 4.00] | 2.00 [0.00 to 12.00] | 2.40 [0.00 to 7.20] | 2.00 [0.00 to 8.00]
Statistical Analysis 1: Comparison: Group I: Placebo vs Group II: Ustekinumab 27 mg Every 4 Weeks vs Group III: Ustekinumab 90 mg Every 8 Weeks vs Group IV: Ustekinumab 90 mg Every 4 Weeks vs Group V: Ustekinumab 180 mg Every 4 Weeks; Hypothesis: The null hypothesis of no effect among the treatment groups was tested against the alternative hypothesis that the cumulative number of newly Gd-enhancing T1-weighted lesions on cranial MRIs through Week 23 would decrease monotonically with dose at a significance level of 0.05; Test type: Superiority or Other; p = 0.00, Jonckheere Terpstra — The p-value was non estimable because the observed trend was in the opposite direction of that stated in the one sided alternative hypothesis; Jonckheere Terpstra nonparametric trend test procedure with 5% level of significance was be used to test for the monotonic trend

2. Secondary Outcome: Relapses of Multiple Sclerosis (MS) Through Week 23
Description: Clinical relapse of MS is defined as any acute neurological event, reported by the patient, that is characterized by new or worsening signs or symptoms of MS lasting at least 48 hours after a stable period of at least 30 days that is considered, in the judgment of the study physician (treating neurologist), to be a clinical relapse of MS.
Time Frame: Week 23
Population: Missing data remained missing. No treatment failure rule was implemented.
Measure: Median (Inter-Quartile Range); unit: Relapses
Arm/Group | Group I: Placebo | Group II: Ustekinumab 27 mg Every 4 Weeks | Group III: Ustekinumab 90 mg Every 8 Weeks | Group IV: Ustekinumab 90 mg Every 4 Weeks | Group V: Ustekinumab 180 mg Every 4 Weeks
Number analyzed (Participants) | 49 | 50 | 50 | 50 | 50
Relapses | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 1.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
Statistical Analysis 1: Comparison: Group I: Placebo vs Group V: Ustekinumab 180 mg Every 4 Weeks; Test type: Superiority or Other; p = 0.892, 2-sided Wilcoxon Mann-Whitney
Statistical Analysis 2: Comparison: Group I: Placebo vs Group IV: Ustekinumab 90 mg Every 4 Weeks; Test type: Superiority or Other; p = 0.599, 2-sided Wilcoxon Mann-Whitney
Statistical Analysis 3: Comparison: Group I: Placebo vs Group III: Ustekinumab 90 mg Every 8 Weeks; Test type: Superiority or Other; p = 0.517, 2-sided Wilcoxon Mann-Whitney
Statistical Analysis 4: Comparison: Group I: Placebo vs Group II: Ustekinumab 27 mg Every 4 Weeks; Hypothesis: The null hypothesis is no difference between any ustekinumab treatment groups and placebo at a significant level of 0.05 for comparison for each treatment group; Test type: Superiority or Other; p = 0.967, 2-sided Wilcoxon Mann-Whitney

3. Secondary Outcome: Change From Baseline in Expanded Disability Status Scale (EDSS)
Description: The EDSS is based on an independent neurologist's examination of 8 functional systems and is used to classify multiple sclerosis (MS) severity, progression, disability, and evaluate treatment results. A numeric score ranging from 0 (normal) to 10 (death) is produced, the change from baseline of the EDSS score ranges from -9 to 10.
Time Frame: Baseline, Week 23
Population: Intent to treat. Missing data was imputed. Missing EDSS scores was replaced with the last non-missing EDSS value observed (last observation carried forward).
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Group I: Placebo | Group II: Ustekinumab 27 mg Every 4 Weeks | Group III: Ustekinumab 90 mg Every 8 Weeks | Group IV: Ustekinumab 90 mg Every 4 Weeks | Group V: Ustekinumab 180 mg Every 4 Weeks
Number analyzed (Participants) | 49 | 50 | 50 | 50 | 50
Units on a scale | 0.00 [-0.50 to 0.00] | 0.00 [-0.50 to 0.00] | 0.00 [0.00 to 0.50] | 0.00 [-0.50 to 0.50] | 0.00 [0.00 to 0.00]
Statistical Analysis 1: Comparison: Group I: Placebo vs Group II: Ustekinumab 27 mg Every 4 Weeks; Test type: Superiority or Other; p = 0.720, Wilcoxon (Mann-Whitney); 2-sided Wilcoxon Mann-Whitney test (α = 0.05) used for each comparison with placebo
Statistical Analysis 2: Comparison: Group I: Placebo vs Group III: Ustekinumab 90 mg Every 8 Weeks; Test type: Superiority or Other; p = 0.152, Wilcoxon (Mann-Whitney); 2-sided Wilcoxon Mann-Whitney test (α = 0.05) used for each comparison with placebo
Statistical Analysis 3: Comparison: Group I: Placebo vs Group IV: Ustekinumab 90 mg Every 4 Weeks; Test type: Superiority or Other; p = 0.431, Wilcoxon (Mann-Whitney); 2-sided Wilcoxon Mann-Whitney test (α = 0.05) used for each comparison with placebo
Statistical Analysis 4: Comparison: Group I: Placebo vs Group V: Ustekinumab 180 mg Every 4 Weeks; Hypothesis: The null hypothesis is no difference between any ustekinumab treatment groups and placebo at a significant level of 0.05 for comparison for each treatment group with placebo; Test type: Superiority or Other; p = 0.292, Wilcoxon (Mann-Whitney); 2-sided Wilcoxon Mann-Whitney test (α = 0.05) used for each comparison with placebo

ADVERSE EVENTS:
Time Frame: 71 weeks
Description: Number of participants in each of the 5 dosage groups in the "Participant Flow" rows is different from number of participants analyzed for safety as the actual dosage of medication received by participants in the 5 groups was different due to unavailability of the study medication
Arm/Group | Group I: Placebo | Group II: Ustekinumab 27 mg Every 4 Weeks | Group III: Ustekinumab 90 mg Every 8 Weeks | Group IV: Ustekinumab 90 mg Every 4 Weeks | Group V: Ustekinumab 180 mg Every 4 Weeks
Serious Adverse Events (participants affected / at risk) | 1/49 | 3/51 | 0/47 | 2/52 | 1/50
Other Adverse Events (participants affected / at risk) | 31/49 | 35/51 | 34/47 | 38/52 | 44/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group I: Placebo (N=49) | Group II: Ustekinumab 27 mg Every 4 Weeks (N=51) | Group III: Ustekinumab 90 mg Every 8 Weeks (N=47) | Group IV: Ustekinumab 90 mg Every 4 Weeks (N=52) | Group V: Ustekinumab 180 mg Every 4 Weeks (N=50)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 1 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group I: Placebo (N=49) | Group II: Ustekinumab 27 mg Every 4 Weeks (N=51) | Group III: Ustekinumab 90 mg Every 8 Weeks (N=47) | Group IV: Ustekinumab 90 mg Every 4 Weeks (N=52) | Group V: Ustekinumab 180 mg Every 4 Weeks (N=50)
Upper respiratory tract infection (Infections and infestations) | 6 | 6 | 8 | 6 | 5
Nasopharyngitis (Infections and infestations) | 5 | 6 | 5 | 5 | 7
Urinary tract infection (Infections and infestations) | 4 | 2 | 2 | 2 | 5
Viral infection (Infections and infestations) | 3 | 2 | 6 | 2 | 1
Influenza (Infections and infestations) | 0 | 2 | 2 | 5 | 1
Sinusitis (Infections and infestations) | 3 | 4 | 0 | 1 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 3 | 0 | 2 | 0
Herpes simplex (Infections and infestations) | 3 | 0 | 3 | 1 | 0
Rhinitis (Infections and infestations) | 3 | 0 | 0 | 0 | 4
Vulvovaginal mycotic infection (Infections and infestations) | 3 | 0 | 0 | 0 | 1
Injection site erythema (General disorders) | 4 | 6 | 6 | 11 | 22
Fatigue (General disorders) | 1 | 8 | 6 | 6 | 6
Injection site pain (General disorders) | 2 | 0 | 2 | 4 | 7
Injection site rash (General disorders) | 1 | 1 | 2 | 3 | 3
Injection site pruritus (General disorders) | 0 | 1 | 0 | 2 | 5
Injection site bruising (General disorders) | 0 | 1 | 0 | 2 | 4
Pain (General disorders) | 0 | 0 | 1 | 1 | 3
Pyrexia (General disorders) | 3 | 1 | 0 | 2 | 1
Chills (General disorders) | 0 | 0 | 0 | 3 | 0
Headache (Nervous system disorders) | 2 | 7 | 5 | 9 | 7
Dizziness (Nervous system disorders) | 1 | 2 | 3 | 2 | 1
Hypoaesthesia (Nervous system disorders) | 3 | 2 | 3 | 1 | 2
Paraesthesia (Nervous system disorders) | 4 | 1 | 2 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 4 | 3 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 4 | 1 | 3 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 1 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 2 | 2 | 1 | 1
Shoulder pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 2 | 1 | 0
Nausea (Gastrointestinal disorders) | 5 | 1 | 2 | 4 | 6
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 2 | 1 | 3
Vomiting (Gastrointestinal disorders) | 1 | 4 | 2 | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 4 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 2 | 3 | 1
Depression (Psychiatric disorders) | 5 | 2 | 2 | 4 | 2
Insomnia (Psychiatric disorders) | 1 | 2 | 1 | 1 | 3
Vertigo (Ear and labyrinth disorders) | 0 | 2 | 1 | 4 | 3
Vision blurred (Eye disorders) | 3 | 0 | 0 | 2 | 3
Eye pain (Eye disorders) | 0 | 0 | 1 | 0 | 3
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 5
Skin laceration (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 3
Hypertension (Vascular disorders) | 1 | 0 | 1 | 3 | 1

LIMITATIONS AND CAVEATS:
The count of patients with any nonserious adverse events (NAE) excludes patients who only had NAE that occurred in <=5% of patients. This information may vary from existing approved labeling and publications due to the requirement of this website.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, the only disclosure restriction on the PI is that the sponsor has 60 days to review results communications prior to public release and can embargo communications regarding trial results for a period that does not exceed 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.